CLINICAL TRIAL: NCT06459843
Title: Combined Effects Of of Pursed Lip Breathing and Coordinated Breathing During Aerobic Exercise on Aerobic Capacity, Dyspnea and Anxiety Level in Adult Patients With COPD
Brief Title: Effects Of of Pursed Lip Breathing and Coordinated Breathing in Adult Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0366
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Aerobic capacity; Coordinated breathing technique; Pursed lip breathing technique.
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pursed lip breathing techniques (Experimental): Pursed lip breathing with aerobic exercise for 4 times per week for 4 week and duration will be 45-60 min. Relax your neck and shoulder muscles. For the use of PLB exercise, the intervention will be given every day till the patient discharged from hospital. Patient will perform 5 sets
  Interventions: Other: pursed lip breathing techniques
- coordinated breathing technique (Active Comparator): The intervention will be given un every day till the patient discharge from hospital. Coordinated breathing with aerobic exercise for 4 times per week for 4 weeks. And duration will be 45-60 min
  Interventions: Other: coordinated breathing technique

INTERVENTIONS:
Other: pursed lip breathing techniques — Relax your neck and shoulder muscles. For the use of PLB exercise, the intervention will be given every day till the patient discharged from hospital. Patient will perform 5 sets. In each set, 10 times will be included. Then, instruct the patient to take deep breath through nose for two counts, and keep mouth closed. Inhale for 2 seconds. Now, ask the patient to purse the lips as if the patient was going to gently flicker the flame of candle. Now the patient will breathe out gently while counting for 4 seconds.
  Arms: pursed lip breathing techniques
Other: coordinated breathing technique — Put one hand on your abdomen. Make your abdomen push out while you breathe in through your nose. Suck in your abdominal muscles. Breathe out using the pursed-lip technique. You should feel your abdomen go down. Repeat three times and rest for two minutes.
  Arms: coordinated breathing technique

SUMMARY:
COPD is the chronic lung condition characterized by the damage and enlargement of the air sacs in the lungs, leading to breathing difficulties. A blockage may develop, which traps air inside your lungs. The patient shows clinical manifestation of cough, wheezing, chest tightness, shortness of breath. This research of randomized clinical trial will check the combined effects of pursed lip breathing and coordinated breathing techniques to improve aerobic capacity and dyspnea in patients with COPD by taking sample of 54 patients through convenience sampling and randomly allocating them to two groups A and B out of which A will receive pursed lip breathing with aerobic exercise for 4 times per week for 4 week and duration will be 45-60 min, B will receive coordinated breathing with aerobic exercise for 4 times per week for 4 weeks. And duration will be 45-60 min.Pre and post training outcomes of aerobic capacity and dyspnea will be measured through Six minute walk test and dyspnea Borg scale, and Saint George respiratory questionnaire. The data will be analyzed through SPSS 21.

ELIGIBILITY:
Inclusion Criteria:

* Age range 25 -45 years(5)
* Adult patient diagnosed with (chronic obstructive pulmonary disease) based on clinical and diagnostic criteria.
* Patient willing and able to participate in an pursed lip breathing and coordinated breathing exercise program
* Gender both male and female

Exclusion Criteria:

* Those who cognitive impairment that might affect their ability to comprehend and follow instructions
* Any contraindication to the use of pursed lip breathing or coordinated breathing exercise as determined by the health care provider.
* Individual with severe musculoskeletal limitations or other physical condition that may hinder the ability to perform exercise
* Individual who have experienced the recent exacerbation of COPD symptoms within past three month

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Six minute walk test | baseline and fourth week
  Patients were instructed to walk back and forth at their own pace in a 35 m corridor. A physiotherapist supervised the test through the course, telling the patient the remaining exercise time every 2 min
Borg dyspnea scale | baseline and fourth week
  Dyspnea during the test was evaluated with the modified Borg dyspnea score. Pulmonary function test, inspiratory capacity, and dyspnea score, together with the walking distance were recorded before and after walking. Modified Borg scale is valid patient self-report scale for measuring breathlessness after exercise with the scaling from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Afzal, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Jinnah Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thurlbeck WM, Muller NL. Emphysema: definition, imaging, and quantification. AJR Am J Roentgenol. 1994 Nov;163(5):1017-25. doi: 10.2214/ajr.163.5.7976869.
- [Background] Rodrigues A, Munoz Castro G, Jacome C, Langer D, Parry SM, Burtin C. Current developments and future directions in respiratory physiotherapy. Eur Respir Rev. 2020 Dec 15;29(158):200264. doi: 10.1183/16000617.0264-2020. Print 2020 Dec 31. PMID 33328280